CLINICAL TRIAL: NCT05711797
Title: An Open, Parallel Study Evaluating the Pharmacokinetic Profile, Safety, and Tolerability of a Single Oral Dose of ZX-7101A Tablets in Subjects with Mild or Moderate Liver Insufficiency and Healthy Subjects
Brief Title: Pharmacokinetic Characteristics of Subjects with Hepatic Insufficiency and Healthy Subjects
Acronym: ZX-7101A-203
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Nanjing Zenshine Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ZX-7101A-203
Record Dates: First submitted 2023-01-16; First posted 2023-02-03 (Actual); Last update posted 2024-11-05 (Actual); Status verified 2024-11

CONDITIONS: Influenza, Human
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Intervention Model Description: 80mg ZX-7101A
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ZX-7101A 80mg Mild or moderate liver insufficiency (Experimental)
  Interventions: Drug: ZX-7101A 80mg
- ZX-7101A 80mg Normal liver function (Experimental)
  Interventions: Drug: ZX-7101A 80mg

INTERVENTIONS:
Drug: ZX-7101A 80mg — ZX-7101A a drug to treatment influenza in Chinese adults

SUMMARY:
The objective of this multicenter, open, single-dose, parallel controlled, Phase I clinical study is to Evaluate a single oral ZX-7101A PK in subjects with varying degrees of (mild or moderate) liver insufficiency compared with healthy subjects matched by age, weight, and sex. And to evaluate the the safety and tolerability of ZX-7101A by a single oral dose in subjects.

The main questions it aims to answer are:

* Evaluate a single oral ZX-7101A PK in subjects with varying degrees of (mild or moderate) liver dysfunction and healthy subjects with normal liver function matched for age, weight, and sex.
* To evaluate the safety and tolerability of ZX-7101A by a single oral dose in subjects.

ELIGIBILITY:
Inclusion Criteria:

* The presence of cirrhosis was confirmed by CT, magnetic resonance imaging (MRI), liver biopsy or noninvasive hepatic fibrosis test.
* The subject was determined to have liver insufficiency based on A Grade A or B on the Child-Pugh scale.
* If the subject has hepatic encephalopathy, the investigator determines that the current condition will not interfere with the subject's ability to provide appropriate informed consent.

Exclusion Criteria:

* Previous or present history of respiratory, blood, cardiovascular, digestive, urinary, endocrine and metabolic, neurological or psychiatric disorders with clinical manifestations.
* People with an allergic disposition (multiple drug and food allergies) or who, as determined by the investigator, are likely to be allergic to the investigational drug product or any component of the investigational drug product.
* A history of gastrointestinal surgery or excision may interfere with oral drug absorption and/or excretion
* Patients with abnormal vital signs at screening visit and baseline visit: ear temperature > 37.5℃, pulse rate > 100 beats/min or < 50 beats/min, systolic blood pressure ≥140 mmHg or < 90 mmHg, diastolic blood pressure ≥90 mmHg or < 50mmHg.
* Participated in clinical studies of any drug or medical device within 3 months prior to screening, and participated in clinical studies of drug for 3 or more times within the last year.
* Severe infection, trauma, or major surgery within 4 weeks prior to screening, or clinically significant (as determined by the investigator) acute illness such as gastrointestinal disease, infection (e.g. respiratory or central nervous system infection, and idiopathic peritonitis) within 2 weeks prior to screening.
* Had used any prescription drugs, Chinese herbs, or over-the-counter drugs (except birth control pills, acetaminophen, and topical over-the-counter preparations) in the 2 weeks prior to enrollment; Unless the principal investigator (PI) and the sponsor agree that the drug used has no impact on the safety and PK results of the study; If the combined drug has a longer half-life (more than 3 days), the required time interval will be longer and should be at least 5 half-lives of the drug.
* Smoking averaged more than 5 cigarettes per day in the 3 months prior to screening, or could not stop using any tobacco products during the study period.
* Persons who consumed more than 14 units of alcohol per week (1 unit = 360mL beer, 150 mL wine or 45 mL 40% spirits) in the 3 months prior to the screening period, or who had a positive alcohol breath test (screening period or baseline period), or who could not abstain during the study period.
* Test positive for hepatitis B (HBV) surface antigen, hepatitis C virus (HCV) antibody, anti-human immunodeficiency virus (HIV) antibody or treponema pallidum antibody.
* Subjects with a history of substance abuse (e.g., morphine, dimethyldioxyamphetamine, methylamphetamine, tetrahydrocannabinol, ketamine, cocaine) or who screened positive for substance abuse.
* Those who received the vaccine within 30 days prior to administration or who planned to receive the vaccine during the study period.
* Donors who donated > 400 mL within 3 months prior to the screening period or > 200 mL within 4 weeks or planned to donate blood during the study period.
* Patients with difficulty in venous blood collection.
* Vigorous exercise should not be prohibited within 48 hours before and during the study period.
* It is expected that patients may be scheduled for surgery or hospitalization during the study.
* Any other circumstances which, in the opinion of the investigator, may affect the subject's ability to provide informed consent or to follow the protocol of the study, to complete the study in accordance with the study procedure, or the subject's participation in the study may affect the results of the study or his or her own safety.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2023-04-12 (Actual); Primary Completion 2024-02-06 (Actual); Study Completion 2024-08-09 (Actual)

PRIMARY OUTCOMES:
Cmax | From dosing to 15 days after medication
  To evaluate the peak concentration of ZX-7101A after a single oral administration in subjects with mild and moderate hepatic insufficiency
AUC | From dosing to 15 days after medication
  To evaluate the area under curve of ZX-7101A after a single oral administration in subjects with mild and moderate hepatic insufficiency

SECONDARY OUTCOMES:
Number of Participants with Treatment-Related Adverse Events as Assessed by CTCAE v5.0 after a single oral administration ZX-7101A | From dosing to 29 days after medication
  The Number of Participants with Treatment-Related Adverse Events will be evaluated as the change of vital signs, electrocardiogram (P Wave, QRS Complex, QT Interval), physical examination, and Laboratory test compared with the baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Xian yu huang, doctor, Study Director — Huashan Hospital
Locations (1):
- Shuguang Hospital, Shanghai University of Traditional Chinese Medicine, Shanghai, China

IPD SHARING:
Plan to Share IPD: No